CLINICAL TRIAL: NCT00754299
Title: Outcome of a Prospective Protocol for Smoking Cessation in Nonunion, Malunion, Osseous Infection, and Infected Nonunion Patients
Brief Title: Smoking Cessation in Nonunion, Malunion, Osseous Infection
Acronym: nicotine
Status: Withdrawn | Type: Observational
Why Stopped: Study could not get funding; research never initiated.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, J. Spence Reid, Principal Investigator, Milton S. Hershey Medical Center
Other Study IDs: 28862
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Fracture Nonunion; Infection
Keywords: nonunion/malunion osseous fractures; nicotine dependent; chronic osseous infection; infected osseous nonunions; Fracture nonunion or infection
MeSH Terms: conditions — Fractures, Ununited; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Study Investigators have seen high rates of tobacco cessation success combining Chantix with the risk of no surgery, should tobacco use continue. Once patients achieve tobacco cessation and undergo surgery, the investigators have seen high rates of union and/or infection resolution. The investigators are looking to document and publish these observations. To date, no studies have been published that have examined the effects of this type of protocol on short and long-term tobacco cessation.

The investigators want to examine and report the outcome of Hershey Medical Center's Orthopaedic Trauma Division's protocol for two endpoints: 1) pre-op tobacco cessation and 2) duration of tobacco cessation. This protocol involves counseling, Chantix, and a 'no-surgery' risk. Patients will be followed postoperatively for success and duration of tobacco cessation, as well as for fracture union and/or infection eradication.

DETAILED DESCRIPTION:
The Study Investigators have a Trauma subspecialty within Orthopaedic Surgery. We take care of numerous patients with ununited or malunited fractures i.e., nonunion/malunion patients, as well as patients with chronic bone infections, and patients with infected nonunions. The literature is replete with articles documenting the negative effects of nicotine on fracture healing and chronic bone infection resolution.(5) Many of our chronic infection and nonunion/malunion patients use nicotine in some form. Most of these patients need additional elective surgery to attain fracture union and/or infection resolution. Thus, we are faced with the dilemma of adding an additional procedure to a patient with proven risk factors for nonunion and continued infection. Much time is spent in clinic counseling patients about smoking cessation, requisite for a successful surgical outcome. Since nicotine is extremely addictive, our efforts at helping our trauma patients relinquish tobacco are not always successful. Many of our patients need pharmacologic help with the goal of cessation, and we have been providing Chantix prescriptions to them. In addition to providing Chantix, we currently present to our patients, as standard of care, a requirement that smoking cessation is necessary prior to performing additional surgical procedures.

Chantix (generic name, varenicline)is a relatively new drug designed for helping with tobacco cessation. It has shown great promise for success since it both decreases cravings for nicotine (the highly addictive active ingredient in tobacco) and diminishes withdrawal symptoms of nicotine. This novel, dual approach works by binding to nicotinic receptors in the brain as a partial agonist, decreasing the pleasurable effects of cigarettes and other tobacco products. Once bound to these receptors, Chantix blocks actual nicotine. While blocking nicotine receptors, it also acts like a weak substitute for nicotine, decreasing symptoms of withdrawal. (2)

Our study will include 60 tobacco-using patients of all ages above 18 with osseous nonunion, malunion, established bone infection, or combined diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a tobacco user and have an osseous nonunion, malunion, infection, or infected nonunion of the Clavicle, Humerus, Radius, Ulna, Pelvis, Femur, Tibia, Fibula, or Calcaneus.
* Subjects must be above age 18, be able to understand and give consent, and be non-pregnant.

Exclusion Criteria:

* Patients unable to understand the protocol, patients allergic to chantix, prisoners, and pregnant patients will be excluded, and patients with pre-existing psychiatric illness.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study will include 60 tobacco-using patients of all ages above 18 with osseous nonunion, malunion, established bone infection, or combined diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Union will be defined as no or minimal pain at the fracture site with direct palpation and weight-bearing when applicable; and radiographically, as a minimum of 3 bridging cortices across the fracture site in anteroposterior, lateral, oblique views. | 24 months

SECONDARY OUTCOMES:
Absence of infection will be assessed by lab values, wound inspection, and radiographic evaluation where indicated. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Spence Reid, MD, Principal Investigator — Penn State Milton S. Hershey Medica Center
Locations (1):
- The Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Porter SE, Hanley EN Jr. The musculoskeletal effects of smoking. J Am Acad Orthop Surg. 2001 Jan-Feb;9(1):9-17. doi: 10.5435/00124635-200101000-00002. PMID 11174159
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Tobin ML. Why choose varenicline (chantix) for smoking cessation treatment? Issues Ment Health Nurs. 2007 Jun;28(6):663-7. doi: 10.1080/01612840701354661. No abstract available. PMID 17613164
- [Background] Varenicline (CHANTIX): a stop-smoking pill. ORL Head Neck Nurs. 2006 Fall;24(4):18-9. PMID 17390707
- [Background] Varenicline (Chantix) for tobacco dependence. Med Lett Drugs Ther. 2006 Aug 14-28;48(1241-1242):66-8. No abstract available. PMID 16977281
- [Background] Gaston MS, Simpson AH. Inhibition of fracture healing. J Bone Joint Surg Br. 2007 Dec;89(12):1553-60. doi: 10.1302/0301-620X.89B12.19671. PMID 18057352